CLINICAL TRIAL: NCT06795529
Title: Randomized Trial of a Targeted Palliative Care Intervention for Patients With Metastatic Breast Cancer
Brief Title: Targeted Palliative Care Intervention for Patients With Metastatic Breast Cancer
Acronym: TARGET-PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Duke University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Co-Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24-723; R01CA299956 (NIH)
Record Dates: First submitted 2025-01-18; First posted 2025-01-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer
Keywords: palliative care; communication about care preferences
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative Care Intervention, "TARGET-PC" (Experimental): Patients randomly assigned to TARGET-PC will receive the palliative care intervention in addition to usual oncology care. Palliative care intervention visits will be conducted by a palliative care physician or advanced practice provider either in-person or with hospital-approved videoconference technology. Patients will be scheduled for their first palliative care visit within four weeks of randomization. Subsequent palliative care intervention visits will be scheduled every four weeks until the patient completes visit five. If a patient cannot be scheduled for intervention visits within four weeks, the palliative care clinician will contact them via telephone within four weeks of their prior contact to maintain their relationship and rapport. Palliative care clinicians will be permitted to conduct an intervention visit over the phone or video if they feel it is appropriate based on the patient's health status.
  Interventions: Other: Palliative Care Intervention, "TARGET-PC"
- Enhanced Usual Care (Active Comparator): The oncology clinicians (physicians and advanced practice providers) of patients randomly assigned to the enhanced usual care condition will receive electronic prompts, encouraging them to discuss and document their patient's care preferences for up to five months after the patient is randomized. The prompts will be sent electronically. The research assistant will send the first electronic prompt on the morning of the outpatient oncology appointment immediately following the visit at which the patient provided informed consent for the study. Subsequent electronic prompts will be sent on the morning of outpatient oncology appointments for five months, but no more often than every four weeks.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Palliative Care Intervention, "TARGET-PC" — Palliative care intervention focused on eliciting patients' goals and values to facilitate discussion and documentation of health care preferences.
  Arms: Palliative Care Intervention, "TARGET-PC"
Other: Enhanced Usual Care — Oncology clinicians will receive an electronic message to encourage them to discuss and document their patients' health care preferences.
  Arms: Enhanced Usual Care

SUMMARY:
Many people living with metastatic breast cancer face challenging symptoms and frequent medical visits. At the same time, conversations about personal goals, values, and preferences for care may not always happen as early or as often as patients and families would like. This multi-site study will test the effectiveness of a five-session palliative care program, designed specifically for people with metastatic breast cancer and their caregivers, to strengthen communication with clinicians about what matters most in their care. The study aims to inform how palliative care services can be delivered in a more timely, personalized, and scalable way for people living with advanced cancers who have long disease trajectories, such as metastatic breast cancer.

DETAILED DESCRIPTION:
The diagnosis of metastatic breast cancer can bring many challenges including physical symptoms, treatment side effects, and emotional stress for patients and their families. Palliative care specialists work alongside the oncology team to help patients and families manage symptoms, communicate effectively with their clinicians, and cope with the impact of living with cancer.

Research has shown that when palliative care and oncology teams collaborate closely, patients often experience better symptom relief, clearer communication about their goals and preferences, improved quality of life and mood, and a stronger understanding of their illness. Caregivers also report feeling more supported and less distressed.

The purpose of this research study is to learn whether a personalized palliative care program for people with metastatic breast cancer and their caregivers, called TARGET-PC, can further improve communication, symptom management, coping skills, and understanding of care.

In this study, 400 patients with metastatic breast cancer and their caregivers will be randomly assigned to receive either the TARGET-PC program or enhanced usual care. Enhanced usual care includes an electronic prompt that reminds oncology clinicians to discuss and record each patient's goals and preferences for care. The study will take place at the Massachusetts General Hospital Cancer Center, Penn Abramson Cancer Center, and Duke Cancer Center.

ELIGIBILITY:
Patient Inclusion Criteria:

* age ≥18 years
* diagnosed with metastatic breast cancer
* within 8 weeks of the oncology visit at which they were identified as having an eligible Epic EOL Care Index (≥ 15)
* functioning independently per an Eastern Cooperative Oncology Group performance status ≤2
* receiving their cancer care at one of the participating institutions
* able to complete questionnaires in English or Spanish

Patient Exclusion Criteria:

* received outpatient palliative care visit within the last six months
* enrolled in hospice services
* diagnosed with a comorbid condition that impairs their ability to understand study procedures and/or consent for the trial as per the report of the oncology clinician(s)

Caregiver Inclusion Criteria:

* age ≥18 years
* identified by the patient as a family member or friend who is primarily involved in their care
* able to complete questionnaires in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Documentation of End-of-Life Care Preferences | From date of randomization until date of death or last follow up assessed up to 60 months
  To compare proportions of patients with clinician-documented end-of-life care preferences in the electronic health record by last follow-up time point or date of death between study groups.

SECONDARY OUTCOMES:
Hospice Utilization | From date of randomization until date of death or last follow up assessed up to 60 months
  To compare proportions of patients using hospice services by last follow up time point or death of death between study groups.
Hospice Length of Stay | From date of randomization until date of death or last follow up assessed up to 60 months
  To compare patients' lengths of stay in hospice between study groups among patients who die during study follow up.
Death in the Hospital | From date of randomization until date of death or last follow up assessed up to 60 months
  To compare proportions of patients dying in the hospital between study groups among patients who die during study follow up.
Patient-reported Communication about End-of-Life Care Preferences | From date of randomization until date of death or last follow up assessed up to 60 months
  To compare proportions with patient-reported communication about their end-of-life care preferences between study groups by last follow-up time point or date of death using the Prognosis and Treatment Perceptions Questionnaire (PTPQ). The PTPQ has a single item in which patients indicate whether they have discussed their end-of-life care wishes with their clinicians (scored dichotomously as "yes or no").

OTHER OUTCOMES:
Patient Quality of Life (Functional Assessment of Cancer Therapy-Breast Scale) | 24 Weeks
  To compare patient-reported quality of life per the Functional Assessment of Cancer Therapy-Breast (FACT-B) Scale between study groups at 24 weeks. The FACT-B total scale scores range from 0-148, with higher scores indicating better quality of life.
Patient Psychological Distress (Hospital Anxiety and Depression Scale - HADS) | 24 weeks
  To compare patient-reported anxiety and depression symptoms per the Hospital Anxiety and Depression Scale (HADS) between study groups at 24 weeks. HADS subscale scores range from 0-21, with higher scores indicating worse distress.
Patient Coping (Brief COPE) | 24 weeks
  To compare patient-reported use of approach-oriented and avoidant coping strategies per the Brief-COPE between study groups at 24 weeks. The Brief-COPE approach-oriented subscale scores range from 6-24, and the avoidant subscale scores range from 4-16, with higher scores indicating greater use of each strategy.
Caregiver Quality of Life (Caregiver Oncology QOL Questionnaire) | 24 Weeks
  To compare caregiver-reported quality of life per the Caregiver Oncology Quality-of-Life Questionnaire (CarGOQoL) between study groups at 24 weeks. The CarGOQoL total scale scores range from 0-100, with higher scores indicating better quality of life.
Caregiver Psychological Distress (Hospital Anxiety and Depression Scale - HADS) | 24 weeks
  To compare caregiver-reported anxiety and depression symptoms per the Hospital Anxiety and Depression Scale (HADS) between study groups at 24 weeks. HADS subscale scores range from 0-21, with higher scores indicating worse distress.
Caregiver Coping (Brief COPE) | 24 weeks
  To compare caregiver-reported use of approach-oriented and avoidant coping strategies per the Brief-COPE between study groups at 24 weeks. The Brief-COPE approach-oriented subscale scores range from 6-24, and the avoidant subscale scores range from 4-16, with higher scores indicating greater use of each strategy.
Caregiver-reported Communication about the Patient's End-of-Life Care Preferences | From date of randomization until date of death or last follow up assessed up to 60 months
  To compare caregiver-reported communication about the patient's end-of-life care preferences between study groups by last follow-up time point or the patient's date of death using the Prognosis and Treatment Perceptions Questionnaire (PTPQ). The PTPQ has a single item in which caregivers indicate whether they have discussed the patient's end-of-life care wishes with their clinicians (scored dichotomously as "yes or no").
Caregiver After Death Assessment | From date of randomization until three months after the patient's death assessed up to 60 months
  To compare caregiver-reported assessment of the patient's end-of-life experiences between study groups among caregivers of patients who die during the study period as measured by three items ranging from 0-10, with higher scores indicating worse quality of end-of-life.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The total scale, subscale scores, and item-level scores from the self-report measures, sociodemographic information, electronic health record data, and palliative care visit surveys will be preserved and stored within a secure computing environment. All participant identifiers will be removed and maintained in a separate secure file that will not be shared to protect confidentiality.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be submitted to a publicly available database within three months of study completion and maintained in perpetuity.
Access Criteria: Most of the scientific data generated in this study, including the self-report and electronic health record data, will be made publicly available through the Harvard Dataverse. However, certain sociodemographic information and any other variables that are considered Protected Health Information and potentially identifying the patient participants (e.g., dates of birth and death) will be restricted. Restricted data would only be made available to users who demonstrate a valid research need and meet conditions of use. In accordance with the data repository methods, we will require the completion of a data use agreement form that stipulates data sharing under IRB-approved protocols.

REFERENCES:
- [Background] Greer JA, Moy B, El-Jawahri A, Jackson VA, Kamdar M, Jacobsen J, Lindvall C, Shin JA, Rinaldi S, Carlson HA, Sousa A, Gallagher ER, Li Z, Moran S, Ruddy M, Anand MV, Carp JE, Temel JS. Randomized Trial of a Palliative Care Intervention to Improve End-of-Life Care Discussions in Patients With Metastatic Breast Cancer. J Natl Compr Canc Netw. 2022 Feb;20(2):136-143. doi: 10.6004/jnccn.2021.7040. PMID 35130492